CLINICAL TRIAL: NCT04309526
Title: Double-Blind, Placebo-Controlled, Randomized, Ascending Single Oral Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of NCO-48 Fumarate in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of NCO-48 Fumarate in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nucorion Pharmaceuticals, Inc. (Industry)
Collaborators: Ligand Pharmaceuticals (Industry); Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCO48F-01
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NCO-48 Fumarate (Experimental): NCO-48 Fumarate
  Interventions: Drug: NCO-48 Fumarate
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NCO-48 Fumarate — NCO-48 Fumarate
  Arms: NCO-48 Fumarate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the safety and tolerability of single oral doses of NCO-48 Fumarate in healthy subjects. The secondary objectives are to evaluate the pharmacokinetic (PK) profile of NCO-48 Fumarate and its active metabolite, tenofovir (TFV), in healthy subjects following single oral doses and to evaluate the effect of food on the PK of a 30 mg dose of NCO-48 Fumarate in healthy subjects.

DETAILED DESCRIPTION:
This is a first-in-human, double-blind, placebo-controlled, randomized, ascending single oral dose study. NCO-48 Fumarate will be assessed in healthy subjects (6 groups of 8 subjects each). Subjects will receive a single oral dose of NCO-48 Fumarate or placebo capsules in 1 or 2 periods, depending on the dose group, under fasting conditions (unless otherwise indicated) and will be followed for a 1-week observation period. Safety assessments will be performed and NCO-48 Fumarate and TFV PK will be assessed. The planned doses for this study are 2, 10, 30, 60, 120, and 240 mg. Each group of 8 subjects (Groups 1 to 6) will be randomized in a 3:1 ratio to receive either NCO-48 Fumarate or placebo (6 subjects to receive active drug and 2 subjects to receive placebo) as a single dose on Day 1 of Period 1 in the fasted state. A preliminary assessment of food effect will be conducted in Group 3. Subjects in Group 3 will receive study drug in Period 1 under fasted conditions and return after a minimum of 14 days to receive study drug under fed conditions. There will be a Screening Period of up to 30 days. All subjects (Periods 1 and 2) will be observed through the morning of Day 3 (48-hour post-dose assessment). Safety assessments and NCO-48 Fumarate and TFV PK sample collection (blood and urine) will occur during this time. Subjects will be discharged from the study site after the 48 hour assessments and return to the study site on Days 5 and 7 (final visit) for follow-up procedures. After the Day 7 follow-up procedures for each group, evaluation of all safety and tolerability data collected during the period, and evaluation of any available PK data, the dose for the next group of subjects will be determined by the Safety Monitoring Panel (SMP).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects 21 to 65 years of age, inclusive.
2. Female subjects of non-childbearing potential must be surgically sterile or postmenopausal, defined as spontaneous amenorrhea for at least 2 years with follicle-stimulating hormone (FSH) in the post-menopausal range at the Screening Visit.
3. Sexually active female subjects of childbearing potential (ie, ovulating, pre-menopausal, and not surgically sterile) with male partners or sexually active male subjects with female partners must agree to use a medically accepted contraceptive regimen during their participation in the study and for 90 days after the last dose of study drug.
4. Male subjects must agree to abstain from sperm donation through 90 days after administration of the last dose of study drug.
5. Body mass index (BMI) within the range of 18.5 to 30.0 kg/m2, inclusive, and body weight >45 kg.
6. Able to communicate effectively with the study personnel.
7. Generally good health based upon the results of medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG, as judged by the Investigator.
8. Nonsmokers, defined as not having smoked in the past 3 months prior to study drug administration.
9. Willing and able to understand and comply with study procedures and restrictions, including confinement to the study site and consumption of study meals, and provide written informed consent according to institutional and regulatory guidelines.
10. Estimated glomerular filtration rate >60 mL/min/1.73 m2 calculated from serum creatinine using the Chronic Kidney Disease Epidemiology Collaboration formula.

Exclusion Criteria:

1. Females who are pregnant or breastfeeding or planning to become pregnant during the study.
2. History or presence of asthma or other clinically significant pulmonary disease, thyroid disease (hypo- or hyperthyroidism), hepatitis (except for resolved hepatitis A), or other liver disease.
3. Have any disease or condition (medical or surgical) that, in the opinion of the Investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous systems; or other conditions that may interfere with the absorption, distribution, metabolism, or excretion of study drug or would place the subject at increased risk.
4. Liver transaminase levels (aspartate aminotransferase or alanine aminotransferase) >10% of the upper limit of normal, or presence of other abnormal laboratory values which are considered clinically significant at the Screening Visit or admission to study site (Day -1).
5. Positive screening for hepatitis B (hepatitis B surface antigen), hepatitis C (hepatitis C antibody), or HIV (anti-HIV-1/2).
6. Has used any other investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug.
7. Use of any of the following:

   * Prescription drugs, other than topical products without significant systemic absorption, use of thyroid medication or hormone replacement therapy for at least 6 months, and hormonal contraceptives, within 14 days or 5 half lives (whichever is longer) prior to the first dose of study drug.
   * Natural health products should be restricted within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study drug.
   * Over-the-counter products and non-prescription drugs other than topical products without significant systemic absorption and/or hormone replacement therapy, within 7 days prior to the first dose of study drug, with the exception of the use of acetaminophen, which is allowed up to 1 g daily up to 24 hours prior to admission to the study site, then prohibited until after the last protocol-specified blood sample.
   * Depot injection or implant of any drug (other than hormonal contraceptives) within 3 months prior to the first dose of study drug.
   * Substances known to be strong inhibitors or inducers of cytochrome P450 enzymes within 14 days prior to the first dose of study drug through the last study visit.
8. Unwilling to refrain from consumption of alcohol within 48 hours prior to each dose administration and during any inpatient period.
9. Positive urine drug screen, positive alcohol breath test, and/or positive cotinine test at the Screening Visit or upon admission to the study site.
10. History of alcohol abuse within 1 year prior to the Screening Visit or regular use of alcohol within 6 months prior to the Screening Visit.
11. Illicit drug use (use of soft drugs [such as marijuana] within 3 months prior to the Screening Visit or hard drugs within 1 year prior to the Screening Visit), significant mental illness, physical dependence on any opioid, or any history of drug abuse or addiction.
12. Inadequate venous access.
13. Recently donated plasma (500 mL) within 7 days prior to study drug administration.
14. Hemoglobin <128 g/L (males) or <115 g/L (females) and hematocrit <0.36 L/L (males) or <0.32 L/L (females) at the Screening Visit.
15. History of photosensitivity while on medication.
16. Deemed by the Investigator, after reviewing medical and psychiatric history, physical examination, or laboratory tests, to be unsuitable for any other reason that may either place the subject at increased risk during participation or interfere with the interpretation of the study outcomes.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Severity of all Adverse Events graded according to the Common Terminology Criteria for Adverse Events (CTCAE) | 30 days
  An adverse event is defined as any untoward medical occurrence in a clinic investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. The severity of all adverse events will be graded according to the CTCAE version 4.0 from dosing until 30 days post dose.

SECONDARY OUTCOMES:
NCO-48 Fumarate Area Under the Concentration-Time Curve (AUC) | 7 days
  Blood samples are to be collected at designated time points for the determination of the NCO-48 Fumarate AUC
NCO-48 Fumarate Maximum Plasma Concentration (Cmax) | 7 days
  Blood samples are to be collected at designated time points for the determination of the NCO-48 Fumarate Cmax.
TFV Area under the Concentration-Time Curve (AUC) | 7 days
  Blood samples are to be collected at designated time points for the determination of TFV AUC .
TFV Maximum Plasma Concentration (Cmax) | 7 days
  Blood samples are to be collected at designated time points for the determination of the TFV Cmax.

CONTACTS AND LOCATIONS:
Overall Officials: Leela Vrishabhendra, MD, Principal Investigator — Medpace Clinical Pharmacology Unit
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No